CLINICAL TRIAL: NCT03744000
Title: Impact of Immediate Stent Implantation Versus Deferred Stent Implantation on Clinical Outcomes in Patients With Anterior Wall ST-segment Elevation Myocardial Infarction
Brief Title: Deferred Stenting in Patients With Anterior Wall STEMI
Acronym: INNOVATIONCORE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Abbott (Industry); Samjin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Dr. Cheol Woong Yu, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INNOVATION-CORE
Record Dates: First submitted 2018-08-21; First posted 2018-11-16 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Acute Myocardial Infarction With ST Elevation; Anterior Wall Myocardial Infarction
Keywords: STEMI; Deferred stenting; Anterior wall myocardial infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Anterior Wall Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Immediate stenting (Placebo Comparator): Within enrolled patients who agreed to participate in the study, signed informed consent and being satisfied with inclusion and exclusion criteria, stent implantation is done on the initial procedure in immediate stenting group.
  Interventions: Procedure: Immediate stenting
- Deferred stenting (Active Comparator): Within enrolled patients who agreed to participate in the study, signed informed consent and being satisfied with inclusion and exclusion criteria, only TIMI Ⅲ flow achievement is done on the initial procedure and stent implantation is deferred for 3-7 days in the deferred stenting group.
  Interventions: Procedure: Deferred stenting

INTERVENTIONS:
Procedure: Immediate stenting — Abciximab (0.25㎎/㎏) intracoronary injection will be performed to all possible patients after guidewire has passed culprit lesion. Additional manual thrombus aspiration or balloon angioplasty can be performed by operator to achieve TIMI Ⅲ flow. When TIMI Ⅲ flow is achieved after these procedures, patient will be randomized to immediate stenting or deferred stenting group. In immediate stenting group, stenting will be done immediate after achieving TIMI III flow during initial procedure.
  Arms: Immediate stenting
Procedure: Deferred stenting — Abciximab (0.25㎎/㎏) intracoronary injection will be performed to all possible patients after guidewire has passed culprit lesion. Additional manual thrombus aspiration or balloon angioplasty can be performed by operator to achieve TIMI Ⅲ flow. When TIMI Ⅲ flow is achieved after these procedures, patient will be randomized to immediate stenting or deferred stenting group. In deferred stenting group, second stage procedure (stent implantation) will be done at 3 to 7 days after TIMI Ⅲ flow has achieved.
  Arms: Deferred stenting

SUMMARY:
Trial Name) Impact of Immediate SteNt ImplaNtatiOn Versus Deferred Stent ImplAntaTION on Clinical Outcomes in Patients with AnteRior Wall ST-segment Elevation Myocardial Infarction (INNOVATION-CORE)

Objectives) To evaluate the impact of deferred versus immediate stenting in patients with acute ST-segment elevation anterior wall myocardial infarction (STEMI) on

1. the clinical efficacy and safety
2. the microvascular obstruction using Cardiac magnetic resonance (MR)
3. the structural and functional cardiac remodeling using conventional echocardiography and strain imaging
4. the intravascular findings using optical coherence tomography (OCT)

Study Design) A multicenter, prospective, randomized, controlled, open-label clinical trial for anterior wall STEMI patients

Patient Enrollment) 460 patients will be enrolled at 20 centers in South-Korea

Patient Follow-Up) Clinical follow-up will occur at 1, 6, 12 months, 2, 3 years and 5 years. Investigator or designee may conduct follow-up as telephone contacts or office visits.

Primary Endpoint) Composite of all-cause death, hospitalization due to heart failure, recurrent myocardial infarction (MI), target vessel revascularization (TVR) at 2 years.

Secondary Endpoints)

1. Clinical events A. All-cause death B. Cardiac death C. Hospitalization due to heart failure D. Recurrent MI E. TVR F. Stent thrombosis
2. Imaging parameters A. Echocardiographic parameters i. Left ventricle (LV) remodeling index ii. %LV strain iii. Regional wall motion abnormality B. Cardiac MR parameters (optional) i. Infarct size ii. Microvascular obstruction (MVO) size iii. MVO incidence iv. MVO to infarct ratio C. OCT parameters (optional) i. Plaque morphology ii. Lipid index iii. Minimal scaffold area and area stenosis iv. Stent malapposition

DETAILED DESCRIPTION:
1. Study background The main treatment for acute ST segment elevation myocardial infarction due to thrombogenesis and complete occlusion resulting from rupture or erosion of the atherosclerotic plaque in the coronary artery is to rapid open of the coronary artery through the coronary intervention. Infarction-associated epicardial coronary arteries reach Thrombolysis In Myocardial Infarction (TIMI) 3 blood flow in approximately 90% of patients after primary coronary intervention. However, many of these patients had microvascular dysfunction assessed by myocardial brush and ST segment complete response, and only about 35% of these patients achieved ideal reperfusion in which blood flow was smoothly delivered to the myocardium and tissue. A "no-reflow" phenomenon or microvascular obstruction, a serious form of microvascular dysfunction, raises the late mortality rate of patients who underwent reperfusion from 1.9 to 7.1 times. It is also well known that the phenomenon increases the incidence of re-infarction and the size of myocardial infarction and induces left ventricular remodeling after several months.

   To date, two treatment strategies have been proven to be effective in the treatment of distal microvascular embolism, which are manual thrombus aspiration and intracoronary administration of abciximab.

   Recently, the theory that deferred stenting can reduce microvascular obstruction has been suggested. The theoretical basis for the hypothesis is that prolonged antiplatelet therapy and anticoagulation for a deferral period may enable the resolution of the thrombus burden in infarct-related arteries, which is a substrate of distal embolization and subsequent microvascular obstruction. additional rationale is what is called the "vascular cooling down" to avoid mechanical stimulus in the milieu of active inflammation within an infarct-related artery in the early stages of myocardial infarction and prolong exposure to intensive statin therapy before stent implantation.

   Based on this theory, four randomized control trials were published recently, but their results were different. According to the subgroup analysis of the INNOVATION study, in the cases of anterior wall myocardial infarction, deferred stenting strategy reduced not only the infarction size but also the incidence of microvascular obstruction. These findings suggest that the left anterior descending artery has more microvascular bed than the other vessels, and thus the positive result of deferred stenting could be maximized. However, these subgroup analysis results do not have sufficient statistical power to conclude deferred stenting is beneficial in the left anterior wall myocardial infarction, it is important to reaffirm the results with a large randomized control trial exclusively selected for left anterior wall myocardial infarction.

   In this study, we sought to evaluate the impact of deferred versus immediate stenting in patients with acute ST-segment elevation anterior wall myocardial infarction on clinical efficacy and safety.
2. Study objectives The primary objective of this study was to evaluate 1) the clinical efficacy and safety of immediate versus deferred stent implantation in patients with acute ST-segment elevation anterior wall myocardial infarction; 2) the degree of microvascular occlusion reflecting distal microvascular embolization using Cardiac MR and 3) the LV strain using echocardiography.
3. Medical devices and therapeutic agents The medical devices and therapeutic agents to be used in this study are the treatment modalities that have been proven to be beneficial in the treatment and prognosis evaluation of acute ST segment elevation myocardial infarction in general. The stent is a third-generation drug-coated stent, and we intend to unify it as one type (Xience alpine, everolimus eluting coronary stent, Abbott, USA) in order to prevent the difference in results due to differences in stent types.
4. Expected effects of the research The treatment of acute myocardial infarction has been continuously developed not only in the revascularization of the coronary arteries but also in the improvement of microvascular perfusion. In addition to conventional thrombus aspiration, the use of Glycoprotein IIb / IIIa inhibitors such as Abxicimab has been used to improve the therapeutic results. However, it is also true that such treatment methods alone have limitations in the prevention and treatment of microvascular obstruction. Recently, deferred stenting has been attracting attention as a new method to reduce microvascular occlusion. Especially, deferred stenting is expected to have a positive result in left anterior wall MI with high microvascular volume. It is expected to be able to determine the effect of deferred stenting strategy on the incidence of clinical events and improvement of microvascular revascularization in patients with ST elevation anterior wall myocardial infarction through this study.
5. Clinical trial monitoring Monitor personnel designated by the investigator to obtain quality test data will review the clinical trial data at appropriate intervals to ensure accuracy, completeness, and compliance with the protocol. The monitoring personnel can investigate all documents and essential records held by clinical investigators or clinical trial laboratories, including the medical records (office, clinic, and hospital) of the subjects participating in the clinical trial. Clinical investigators and researchers should allow access to these records to the monitoring personnel. The monitoring plan will be conducted three times in total, at the time of registering the number of subjects corresponding to 50% or more of the total enrollment number, when the completed research subject reaches 70% or more, and immediately before the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Typical ischemic chest pain lasting more than 30 minutes
2. New ST elevation at the J point in two contiguous leads with the cut-points: ≥0.1 mV in all leads other than leads V2-V3 where the following cut-points apply: 0.2 ≥mV in men ≥40 years; ≥0.25 mV in men <40 years, or ≥0.15 mV in women27 or new left bundle branch block28.
3. Symptom onset of chest pain within 6 hours
4. If left anterior descending artery is culprit lesion on coronary angiography (Ostium to mid lesion). However, if the right coronary artery is hypoplastic and the distal portion of the left anterior descending artery feeds to the area of the posterior lower coronary artery (PDA), culprit lesion of the distal part of left anterior descending artery can also be included in the study.
5. If TIMI blood flow before intervention is 0, 1 or 2
6. If TIMI 3 blood flow was secured before coronary stenting by intracoronary abciximab injection, manual thrombus aspiration and balloon dilatation
7. Patients who wrote the informed consent: The subject should be able to receive informations of treatment, risks, effects and other therapeutic modalities regarding staged percutaneous coronary intervention (PCI) at least verbally, and investigators should be provided written informed consent from a subject or a legally recognized representative prior to giving any treatment related to the study.

Exclusion Criteria:

1. If there is a previous history of myocardial infarction or coronary artery bypass surgery
2. Cardiogenic shock
3. Rescue PCI after thrombolytic therapy
4. If the life expectancy of the accompanying disease is expected to be less than one year or the patient is not cooperating with the protocol.
5. In cases where the left main lesion is an infarction related artery (If the left main lesion is a simple left main branch lesion rather than an infarction related vessel, it is included in the study)
6. STEMI due to Stent thrombosis
7. A major dissection (Type C to F) occurred during the procedure including balloon dilatation for securing TIMI blood flow and the risk of acute closure at the time of staged stenting was expected

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2025-04-03 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
composite of all-cause death, hospitalization due to heart failure, recurrent MI, TVR, major adverse cardiovascular events (MACE) | Initial admission date to last outpatient clinic visit or clinical outcome of interest occurs, whichever occur first, assessed up to 5 years

SECONDARY OUTCOMES:
All-cause death | Initial admission date to last outpatient clinic visit or clinical outcome of interest occurs, whichever occur first, assessed up to 5 years
Cardiac death | Initial admission date to last outpatient clinic visit or clinical outcome of interest occurs, whichever occur first, assessed up to 5 years
Hospitalization due to heart failure | Initial admission date to last outpatient clinic visit or clinical outcome of interest occurs, whichever occur first, assessed up to 5 years
Recurrent MI | Initial admission date to last outpatient clinic visit or clinical outcome of interest occurs, whichever occur first, assessed up to 5 years
TVR | Initial admission date to last outpatient clinic visit or clinical outcome of interest occurs, whichever occur first, assessed up to 5 years
Stent thrombosis | Initial admission date to last outpatient clinic visit or clinical outcome of interest occurs, whichever occur first, assessed up to 5 years
MVO volume | Post MI 30 days
MVO incidence | Post MI 30 days
MVO to infarct size | Post MI 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Woong Yu, M.D.,Ph.D., Principal Investigator — Cardiovascular center, Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided